CLINICAL TRIAL: NCT01081366
Title: Evaluation of the Safety Profile of the Pantera Lux Paclitaxel Releasing Balloon for Coronary Arteries in Daily Clinical Practice
Brief Title: Drug Eluting Pantera Lux Catheter Registry
Status: Completed | Type: Observational
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Other Study IDs: C0905 DELUX
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
All comers registry - Evaluation of the safety and efficacy of the Pantera Lux Paclitaxel releasing balloon for coronary arteries in daily clinical practice.

DETAILED DESCRIPTION:
All patients are treated with the Pantera Lux Paclitaxel releasing balloon.

Clinical follow ups at 1, 6 and 12 months after coronary intervention.

ELIGIBILITY:
Inclusion criteria:

* Signed Patient Informed Consent / Data Release Form
* Patient eligible for percutaneous coronary intervention (PCI)
* Patient is older than 18 years of age

Exclusion Criteria

* Patient has a known allergy against appropriate anticoagulation / antiplatelet therapy
* Patients with known allergy against paclitaxel or BTHC
* Patients with a target lesion that was previously treated by brachytherapy
* Pregnant woman or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All comers registry. Patients treated with the Pantera Lux Paclitaxel releasing balloon catheter are enrolled consecutively to represent a typical set of patients at each site.
Sampling Method: Non-Probability Sample
Enrollment: 1064 (Actual)
Dates: Start 2010-04; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | 6 M
  Death, non-fatal MI, clinically driven target vessel revascularization (TVR)

SECONDARY OUTCOMES:
MACE | 12 M
  Death, non-fatal MI, clinically driven TVR
All MACE | 1, 6, and12 M
  Death, non-fatal MI, any revascularization
Clinically driven TVR | 1, 6 and 12 M
Acute success | Post procedure
  Clinical device success, clinical procedure success

CONTACTS AND LOCATIONS:
Overall Officials: Raph Toelg, MD, Principal Investigator — Herz-Kreislauf-Zentrum, Segeberger Kliniken GmbH, Am Kurpark 1, 23795 Bad Segeberg, Germany
Locations (1):
- Herz-Kreislauf-Zentrum, Segeberger Kliniken GmbH, Bad Segeberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Toelg R, Merkely B, Erglis A, Hoffman S, Bruno H, Kornowski R, Slagboom T, Naber C, Witzenbichler B, Graf K, Richardt G, Hehrlein C; DELUX investigators. Coronary artery treatment with paclitaxel-coated balloon using a BTHC excipient: clinical results of the international real-world DELUX registry. EuroIntervention. 2014 Sep;10(5):591-9. doi: 10.4244/EIJV10I5A102. PMID 24345357